CLINICAL TRIAL: NCT01027819
Title: Comparison of Outcomes in Mobile and Fixed-bearing Total Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNUHOSK09MBFB; SNUHOSK09MBFB (Other: Seoul national university hospital)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Results first posted 2011-04-05 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Osteoarthritis of Knee
Keywords: Total knee arthroplasty; Mobile bearing; Fixed bearing; Range of motion; Knee Society Score
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile bearing (Active Comparator): Mobile bearing type between polyethylene insert and tibial component MB type will be randomly used in total knee arthroplasty
  Interventions: Device: Mobile bearing
- Fixed bearing (Active Comparator): Fixed bearing type between polyethylene insert and tibial component FB type will be randomly used in total knee arthroplasty
  Interventions: Device: Fixed bearing

INTERVENTIONS:
Device: Mobile bearing — Mobile bearing in total knee arthroplasty
  Other Names: Zimmer LPS-flex mobile bearing type polyethylene insert
  Arms: Mobile bearing
Device: Fixed bearing — Fixed bearing in total knee arthroplasty
  Other Names: Zimmer LPS-flex fixed bearing in polyethylene insert
  Arms: Fixed bearing

SUMMARY:
The purpose of this study is to compare the clinical and radiological outcomes of mobile-bearing with that of fixed-bearing in total knee arthroplasty.

DETAILED DESCRIPTION:
Double blind, randomized prospective study Mobile or fixed bearing of the same company

* Mobile bearing group : group M
* Fixed bearing group : group F

Inclusion criteria

* patients expected primary total knee arthroplasty without severe deformity

Clinical outcomes

* Range of motion
* Complication
* Scorings

  * KSS, KSFS, HSS score, WOMAC score, Oxford score, SF-36

Radiological outcomes

* Alignment angles in knee
* Positions of femoral and tibial components
* Position of patella
* Radiolucency

ELIGIBILITY:
Inclusion Criteria:

* primary total knee arthroplasty

Exclusion Criteria:

* infection
* severe deformity in knee
* revision

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-11; Primary Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Myung Chul Lee, M.D., Ph. D., Study Director
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was started from Sep 2005 to Aug 2006 in medical clinic and randomly allocated into two groups.
Groups:
- Mobile Bearing; Fixed Bearing: Mobile bearing vs Fixed bearing
Period: Overall Study
Arm/Group | Mobile Bearing | Fixed Bearing
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Bearing | Fixed Bearing | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 17 | 26
  >=65 years | 31 | 23 | 54
Age Continuous [Mean (Standard Deviation); unit: years] | 68.36 (5.61) | 66.08 (5.55) | 67.24 (5.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 38 | 39 | 77
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Rotational Angle Between Femur and Tibia
Time Frame: 2 weeks
Population: The rotational angle between the femur and tibia was collected by postoperative CT and asssessed between the transepicondylar angle in the femur and the vertical line of the AP axis of the tibia(the line between the insertion of the PCL and the medial 1/3 point of the tibial tuberosity).
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Mobile Bearing | Fixed Bearing
Number analyzed (Participants) | 40 | 40
degree | -0.48 (2.18) | -0.66 (1.52)

2. Secondary Outcome: Knee Society Score
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Mobile Bearing | Fixed Bearing
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
First, our study population is composed of elderly patients with large female dominance

Second concern was inherent errors in making the measurements in this kind of study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No